CLINICAL TRIAL: NCT04439461
Title: Adaptation and First Step Validation of the International Classification of Functioning, Disability and Health Core Set for Vocational Rehabilitation for Cancer Survivors: A Sequential Mixed Method Study
Brief Title: Adaptation and First Step Validation of the ICF Core Set for Vocational Rehabilitation for Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Sara Paltrinieri, MSc Occupational Therapist, Azienda USL Reggio Emilia - IRCCS
Other Study IDs: CS-VR-ONCO_MFR_2020
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Cancer Survivors
Keywords: Vocational Rehabilitation; International Classification of Functioning, Disability and Health; Return to Work

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Return to work (RTW) of cancer survivors (CSs) is an emerging health issue, as cancer incidence, survival rate and prevalent cases have increasing trends and more than 1/3 of CSs are in their working age.

Starting from the International Classification of Functioning, Disability and Health (ICF), the Core Set for Vocational Rehabilitation (CS-VR) has been developed to comprehensively describe work functioning of individuals reporting difficulties and in need of VR. The CS-VR guides the multidisciplinary assessment of individuals and the planning of appropriate VR interventions but, to date, it has been tested only in spinal cord injury and musculoskeletal diseases. Thus, verifying the appropriateness of the CS-VR in a population of cancer survivors seems a step forward.

This sequential mixed method study aims to adapt and validate the CS-VR in Italian cancer survivors, defining the minimum standard of work functioning areas to assess in this population.

DETAILED DESCRIPTION:
Starting from the CS-VR, this study aims to define the CS-VR-Onco, an ICF core set consistent with cancer survivors' needs.

CS-VR-Onco will guide professionals in:

1. comprehensively assessing work functioning
2. identifying the areas of work functioning in which the VR intervention is relevant
3. identifying patients who would benefit most from VR
4. measuring work functioning pre-post VR

This sequential exploratory design involves multiple phases of qualitative (phase 1) and quantitative (phase 2) data collection.

Qualitative_phase 1, To adapt the CS-VR: 1.a_Focus groups (FGs) will be organized with CSs selected from the UNAMANO project (NCT03666936), the Cancer Registry of Reggio Emilia, the General Practitioners of the province of Reggio Emilia and the voluntary non-profit associations of cancer patients. During the FGs, we will ask participants to name and reflect on barriers and facilitators influencing their RTW process. Further, the FGs will address those ICF components from which the CS-VR categories were extracted. 1.b_Consensus-based approach with a sample of stakeholders of the RTW process. We will integrate evidence gathered from phase 1.a and the literature to develop the minimum standard for the assessment of work functioning in this population (CS-VR-Onco).

Quantitative_phase 2, To validate the CS-VR-Onco: 2.a_Cross-sectional survey of CSs extracted from the Cancer Registry of Reggio Emilia. Through a guided interview based on the categories of the CS-VR-Onco, we will ask participants to report their work difficulties. 2.b_Longitudinal study on cancer patients recently diagnosed with cancer referred to UNAMANO project for VR. Before and after the VR, CS-VR-Onco will be administer to identify patients' needs. Additionally, participants will be assessed with valid measurement tools (when present) pertinent to the CS-VR-Onco categories identified.

ELIGIBILITY:
1. Inclusion Criteria:

   * cancer diagnosis
   * CSs employed at diagnosis

   Exclusion Criteria:
   * comorbidities that limit communication or collaboration (i.e., aphasia, dementia, etc.)
   * non-melanoma skin cancer
2. Inclusion Criteria: Stakeholders who handle the RTW process: healthcare professionals, social workers, CSs, caregivers, employers, nonprofit associations, vocational counsellors, etc.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1.a Focus Group: CSs will be recruited if the eligibility criteria reported below are satisfied. The Cancer Registry of Reggio Emilia will recruit CSs diagnosed in 2017 and who have already returned to work. 1.b Consensus-based approach: stakeholders (healthcare professionals, social workers, CSs, caregivers, employers, nonprofit associations, vocational counsellors, etc.) who handle the RTW process of CSs will be invited to participate. 2.a Cross-sectional study: CSs will be recruited if the eligibility criteria reported below are satisfied and diagnosis occurred in 2018. 2.b Longitudinal study: participants will be recruited if the eligibility criteria reported below are satisfied and cancer patients will be referred to UNAMANO for VR.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
1.a_Focus group | 3 months
  To obtain the preliminary CS-VR-Onco, which categories will be subsequently analyzed by the group of stakeholders.
1.b_Consensus-based approach | 3 months
  To obtain the CS-VR-Onco, that is representative of minimum standard of work functioning areas to be assessed in cancer survivors in working age.

SECONDARY OUTCOMES:
2.a_Cross-sectional survey | 12 months
  To describe the frequency of distribution of the categories included in the CS-VR-Onco (content validity) and to compare those distributions between CSs who did and those who did not experience difficulties in the RTW process (construct validity).
2.b_Longitudinal study | 12 months
  To verify whether the CS-VR-Onco can appropriately identify the categories in which VR is of main relevance and detect changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Paltrinieri, Msc OT, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Azienda Unità Sanitaria Locale Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Derived] Paltrinieri S, Costi S, Pellegrini M, Diaz Crescitelli ME, Vicentini M, Mancuso P, Giorgi Rossi P, Fugazzaro S, Mazzini E, Escorpizo R, Ghirotto L. Adaptation of the Core Set for Vocational Rehabilitation for Cancer Survivors: A Qualitative Consensus-Based Study. J Occup Rehabil. 2022 Dec;32(4):718-730. doi: 10.1007/s10926-022-10033-y. Epub 2022 Mar 25. PMID 35334038